CLINICAL TRIAL: NCT01096810
Title: A Phase II Trial of TBL 12 Sea Cucumber Extract in Patients With Untreated Asymptomatic Myeloma
Brief Title: Study of TBL 12 Sea Cucumber Extract for Patients With Untreated Asymptomatic Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The research is permanently closed to enrollment.
Sponsor: Jagannath, Sundar, M.D. (Individual)
Collaborators: Unicorn Pacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBL 12
Record Dates: First submitted 2010-02-22; First posted 2010-03-31 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Myeloma
Keywords: Asymptomatic
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TBL 12 (Experimental): TBL 12, sea cucumber, will be administered orally at a dose of 2 units (20 mL each) twice a day until disease progression
  Interventions: Drug: TBL 12

INTERVENTIONS:
Drug: TBL 12 — TBL 12 will be administered orally at a dose of 2 units (20 mL each) twice a day until disease progression.
  Other Names: Sea Cucumber

SUMMARY:
Purpose:

The purpose of this study is to see if TBL 12, which is a blend of Sea Cucumber, Sea Sponge, Shark Fin, and Sea Urchin (animals that live in the Pacific Ocean) as well as Sargassum (a plant that lives in the Pacific Ocean), will have effects against asymptomatic multiple myeloma and to see what the side effects are.

Eligibility:

Several criteria must be met to be eligible for this study, including but not limited to the following:

* a diagnosis of asymptomatic multiple myeloma
* adequate cardiac, liver and kidney function
* age 18 and older

DETAILED DESCRIPTION:
Multiple myeloma is a cancer that evolves from a state known as Monoclonal Gammopathy of Undetermined Significance (MGUS), defined by parameters of M spike and bone marrow. After evolution to myeloma, patients may be asymptomatic, that is, without any endorgan disease of hypercalcemia, renal insufficiency, anemia or bone lesions. In asymptomatic myeloma (ASxM), there is no standard therapy. Thalidomide has been tried in patients with ASxM but with significant toxicity. The patients with ASxM are evaluable in terms of paraprotein measurements. TBL12 sea cucumber extract has been shown to have a number of antitumor properties preclinically, including antiangiogenesis and direct tumor cytotoxicity. TBL12 has been used by a number of patients as a food supplement without any toxicity detected. We thus propose to determine the clinical activity of this agent in patients with ASxM. Patients will be given TBL12 at the dose of 2 units of 20 mL each twice per day daily for one year and the effects on the paraprotein noted. Clinical effects seen will be correlated with any in vitro changes in angiogenesis in patient bone marrow samples. The results of this trial may form the basis for the use of this nontoxic agent in patients with the prodrome of or with other early cancers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma
* Measurable disease
* For non-secretors, measurable protein by Freelite or plasmacytoma
* Asymptomatic disease

Exclusion Criteria:

* POEMS syndrome
* Plasma cell leukemia
* Receiving steroids greater than the equivalent of 10 mg prednisone
* Infection not controlled by antibiotics
* HIV infection
* Known active hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Jagannath, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TBL 12
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TBL 12
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 58 [22 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 20
Bone Marrow Plasmacytosis [Number; unit: percentage of participants] | 38

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: To determine the time to progression of asymptomatic multiple myeloma patients receiving TBL 12. The time to progression will be measured in units of a cycle (28 day cycles).
  Progression is defined using the International Uniform Response Criteria for Multiple Myeloma (Leukemia (2006)20:1467-1473). Which requires one or more of the following: >25% increase in SPEP (must also be an absolute increase of at least 5 g/dL), >25% increase in UPEP (must also be an absolute increase of at least 200 mg/24 hours), >25% increase in bone marrow plasma cells (must also be an absolute increase of at least 10%), new lytic bone lesions or soft tissue plasmacytomas, or development of hypercalcemia (not attributable to any other cause).
Time Frame: From date of treatment until the date of first documented progression
Measure: Median (Full Range); unit: cycles
Arm/Group | TBL 12
Number analyzed (Participants) | 20
cycles | 15 [2 to 54]

2. Primary Outcome: Response Rate
Description: The response rate - percentage of participants with overall response.
  Overall response for any participants that has achieved at least a PR or better (PR, VGPR, CR, sCR) is defined using the International Uniform Response Criteria for Multiple Myeloma (Leukemia (2006)20:1467-1473) . Which requires the following: at least >50% reduction in SPEP, at least >90% reduction or <200 mg in UPEP, at least >50% reduction in the size of soft tissue plasmacytomas, no lytic bone lesions or similar definition that is accurate and appropriate.
Time Frame: from date of start of treatment until the date of best documented response up to date of progression
Measure: Number; unit: percentage of participants
Arm/Group | TBL 12
Number analyzed (Participants) | 20
percentage of participants | 5

3. Secondary Outcome: Antitumor Effect
Description: To study the possible mechanisms involved in the clinical antitumor effect with determination of inhibition of angiogenesis
Time Frame: Antitumor effect
Population: immunophenotyping was not performed in this study
Arm/Group | TBL 12
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | TBL 12
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBL 12 (N=20)
Pneumococcal Pneumonia (General disorders) | 1 (1) — Pneumococcal pneumonia requiring admission, which was felt to be unrelated to study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBL 12 (N=20)
Nausea (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes